CLINICAL TRIAL: NCT04330924
Title: Nurse-Physician Communication Team Training in Virtual Reality Versus Live Simulations: Randomized Controlled Study
Brief Title: A Comparison Between Physical and Virtual Simulation: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Liaw Sok Ying, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: S-17-107
Record Dates: First submitted 2020-03-26; First posted 2020-04-02 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Interdisciplinary Communication
Keywords: team training; virtual reality; simulation; nurse-physician communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): 3D avatar in a virtual simulation environment
  Interventions: Other: Create Real-life Experience And Teamwork In Virtual Environment (CREATIVE)
- Live Simulation (No Intervention): Live-based simulation in a simulation ward

INTERVENTIONS:
Other: Create Real-life Experience And Teamwork In Virtual Environment (CREATIVE) — 3D virtual hospital environment where participants can perform physical and social interaction and presence using avatars.
  Arms: Virtual Reality

SUMMARY:
Nurse-physician communication skills can be improve through inter-professional team training. Simulation is often used to conduct these training. However, constraints to conduct these sessions such as scheduling and logistic arrangements have been widely reported. Thus with the advancement of technology in education, the use of virtual environment to conduct the team training is being explored and evaluated.

DETAILED DESCRIPTION:
All recruited participants underwent a 3-hour nurse-physician communication training prior to the simulation session. Team Strategies and Tools to Enhance Performance and Patient Safety (TeamSTEPPS) curriculum and pre-learning videos were introduced to the participants. Pre-test questionnaires were administered after the training. Participants were then randomized to the control (live simulation) or intervention group (virtual simulation).

Intervention group participants will undergo a virtual simulation session training via the multi-user virtual world by logging in into the 3D virtual environment while participants in the control group performed the simulations in a physical simulated ward setting. Each pair of 1 medical student and 1 nursing student participate in two role-playing simulation scenarios (15-20 minutes each) along with a facilitator who will provide a debrief (30-minutes). Prior to the simulation, participants were given a smart-watch to monitor their physiological parameters such as heart rate. Post-test questionnaires were administered after the simulation sessions.

After the simulation training, a 30-minutes team-based assessments were conducted based on a inter-professional bedside care scenario in pairs of one medical and one nursing student within their randomized group. The assessments were video recorded for evaluation by assessors who are blinded to the groupings. All participants were then invited to complete a follow-up questionnaire 2 months after the simulation training.

ELIGIBILITY:
Inclusion Criteria:

i) Full time students undertaking National University of Singapore's

* Third or fourth year Bachelor of Science (Nursing)
* Third or fourth year Bachelor of Medicine & Bachelor of Surgery

ii) Completed acute care management modules

Exclusion Criteria:

i) Does not voluntarily agree to join the study

ii) Does not want their performance to be video-recorded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Demographics | Baseline
  Collection of participant demographic data.
Communication skill performance | Post-test (immediately after simulation assessment)
  Participants nurse-doctor communication skill was measured using a validated team communication scale that was self-developed. It is a 7-item checklist with a 5-point scale. The score ranges from 5 to 35 with higher score indicating better nurse-doctor communication performance.
Baseline (Attitudes Toward Interprofessional Health Care Team) | Pre-test
  Measurement of participants' attitudes towards working in interprofessional care team using the 14-item Attitudes Toward Interprofessional Health Care Team questionnaire using a 5-point scale. The scores ranges from 14 to 70 with higher score indicating more positive attitudes.
Post-test (Change of Attitudes Toward Interprofessional Health Care Team from baseline) | Post-test (immediately after simulation training)
  Measurement of participants' attitudes towards working in interprofessional care team using the 14-item Attitudes Toward Interprofessional Health Care Team questionnaire using a 5-point scale. The scores ranges from 14 to 70 with higher score indicating more positive attitudes.
Follow-up (Change of Attitudes Toward Interprofessional Health Care Team from baseline and post-test) | Follow-up (2-months after simulation training)
  Measurement of participants attitudes towards working in interprofessional care team using the 14-item Attitudes Toward Interprofessional Health Care Team questionnaire using a 5-point scale. The scores ranges from 14 to 70 with higher score indicating more positive attitudes.
Baseline (Interprofessional Socialization and Valuing Scale) | Pre-test
  Measurement of participants behaviors, beliefs and attitudes in interprofessional socialization using the 24-item Interprofessional Socialization and Valuing Scale questionnaire using a 7-point scale (1= not at all ; 7= to a very great extent; "not applicable" response is also available). The score ranges from 24 to 168 with higher score indicating greater presence of the attributes measured.
Post-test (Change of Interprofessional Socialization and Valuing Scale from baseline) | Post-test (immediately after simulation training)
  Measurement of participants behaviors, beliefs and attitudes in interprofessional socialization using the 24-item Interprofessional Socialization and Valuing Scale questionnaire using a 7-point scale (1= not at all ; 7= to a very great extent; "not applicable" response is also available). The score ranges from 24 to 168 with higher score indicating greater presence of the attributes measured.
Follow-up (Change of Interprofessional Socialization and Valuing Scale from baseline and post-test) | Follow-up (2-months after simulation training)
  Measurement of participants behaviors, beliefs and attitudes in interprofessional socialization using the 24-item Interprofessional Socialization and Valuing Scale questionnaire using a 7-point scale (1= not at all ; 7= to a very great extent; "not applicable" response is also available). The score ranges from 24 to 168 with higher score indicating greater presence of the attributes measured.
Pulse rate | Pre-test
  Stress measurement parameter using a continuous monitoring smart watch
Pulse rate (Change of parameter from baseline) | Post-test (immediately after simulation training)
  Stress measurement parameter using a continuous monitoring smart watch
Blood pressure (diastolic & systolic) | Pre-test
  Stress measurement parameter using a sphygmomanometer
Blood pressure (diastolic & systolic) (Change of parameter from baseline) | Post-test (immediately after simulation training)
  Stress measurement parameter using a sphygmomanometer
Baseline (State-Trait Anxiety Inventory) | Pre-test
  Measurement of participants state anxiety were measured using the 20-items State-Trait Anxiety Inventory questionnaire using a 4 point likert scale (almost never-almost always). The score ranges from 20 to 80 with higher score indicating higher sense of anxiety.
Post-test (Change of State-Trait Anxiety Inventory from baseline) | Post-test (immediately after simulation training)
  Measurement of participants state anxiety were measured using the 20-items State-Trait Anxiety Inventory questionnaire using a 4 point likert scale (almost never-almost always). The score ranges from 20 to 80 with higher score indicating higher sense of anxiety.
Baseline (Confidence and self-efficacy) | Pre-test
  Measurement of participants confidence and self-efficacy was measured using a 5-items self-efficacy questionnaire through a 10-point likert scale ranging from scores ranging from 5 to 50 with higher score indicating better self-efficacy in their ability in contributing to patient-centered care in a multidisciplinary team.
Post-test (Change of Confidence and self-efficacy from baseline) | Post-test (immediately after simulation training)
  Measurement of participants confidence and self-efficacy was measured using a 5-items self-efficacy questionnaire through a 10-point likert scale ranging from scores ranging from 5 to 50 with higher score indicating better self-efficacy in their ability in contributing to patient-centered care in a multidisciplinary team.
Baseline (Student Stereotype Rating) | Pre-test
  Measurement of participants stereotype towards other health disciplines was measured using the 9-items Student Stereotype Rating Questionnaire through a 5-point Likert scale (1=very low to 5= very high).
  The score ranges from 9 to 45 with higher scores indicating higher perceived ability of the particular healthcare discipline by the other discipline.
Post test (Change of Student Stereotype Rating from baseline) | Post-test (immediately after simulation training)
  Measurement of participants stereotype towards other health disciplines was measured using the 9-items Student Stereotype Rating Questionnaire through a 5-point Likert scale (1=very low to 5= very high). The score ranges from 9 to 45 with higher scores indicating higher perceived ability of the particular healthcare discipline by the other discipline.
Follow up (Change of Student Stereotype Rating from baseline and post test) | Follow-up (2-months after simulation training)
  Measurement of participants stereotype towards other health disciplines was measured using the 9-items Student Stereotype Rating Questionnaire through a 5-point Likert scale (1=very low to 5= very high). The score ranges from 9 to 45 with higher scores indicating higher perceived ability of the particular healthcare discipline by the other discipline.

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liaw SY, Sutini, Chua WL, Tan JZ, Levett-Jones T, Ashokka B, Te Pan TL, Lau ST, Ignacio J. Desktop Virtual Reality Versus Face-to-Face Simulation for Team-Training on Stress Levels and Performance in Clinical Deterioration: a Randomised Controlled Trial. J Gen Intern Med. 2023 Jan;38(1):67-73. doi: 10.1007/s11606-022-07557-7. Epub 2022 May 2. PMID 35501626
- [Derived] Liaw SY, Ooi SW, Rusli KDB, Lau TC, Tam WWS, Chua WL. Nurse-Physician Communication Team Training in Virtual Reality Versus Live Simulations: Randomized Controlled Trial on Team Communication and Teamwork Attitudes. J Med Internet Res. 2020 Apr 8;22(4):e17279. doi: 10.2196/17279. PMID 32267235